CLINICAL TRIAL: NCT05098925
Title: Study of Thermoregulatory Processes in Ultra-endurance Runners in a Hot and Humid Environment
Acronym: ERUPTION-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021/CHU/25
Record Dates: First submitted 2021-09-15; First posted 2021-10-28 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Intensive Sport

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Study of Thermoregulatory Processes in Ultra-endurance Runners in a Hot and Humid Environment
  Interventions: Other: Biological testing

INTERVENTIONS:
Other: Biological testing — Blood sampling, microcapillary sampling, temperature monitoring, saliva testing, EHI questionnaire

SUMMARY:
Human beings are characterized by their extraordinary ability to thermoregulate.

During a physical exercise, only 20% of the energy provided by the substrates is converted into muscular mechanical work. The remaining 80% is released as heat. In temperate environments, so-called metabolic heat is dissipated by several physical phenomena (radiation, conduction, convection and evaporation). However, if the dissipation capacity (in a hot and humid environment for example) is lower than the production of metabolic heat, the body temperature increases progressively until exercise stops or heat-related pathologies develop. This pathological entity defined by the acronym EHI for Exertional Heat Illness gather a wide spectrum of clinical forms ranging from oedema or heat rash, to muscle cramps, to syncope; up to more serious forms such as heat exhaustion or heat stroke during exercise.

Heatstroke during exercise is the second most common cause of death in athletes after heart disease.

However, the results of the epidemiological studies and the recommendations are limited to events with effort durations or distances not exceeding those of the marathon. They therefore do not consider ultra-endurance disciplines.

These disciplines, defined by durations of effort of at least 6 hours, have specific characteristics (duration of effort, intensity, steep gradients, exotic destinations, extreme environments) which means that extrapolation of the results and knowledge of the physiology of thermoregulation from "classic" endurance events, such as marathons, to ultra-endurance events is hazardous. There are therefore significant areas of uncertainty in understanding the thermoregulatory function, prevalence of EHI (Exertional Heat Illness) and health implications of ultra-endurance running in a hot environment. This is the context of ERUPTION-2.

ELIGIBILITY:
Inclusion Criteria:

* Runners participating in " La diagonale des fous " race of the "Grand Raid" 2021 on Reunion Island

Exclusion Criteria:

* Runners who do not understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Core temperature measurement | during 3 days of the race
  Measure of core temperature (°C) will be carried out by continuous monitoring using e-Celsius performance Bodycap technology sensors carried by the athletes through the race
Natremia measurement | during 3 days of the race
  Measure of natremia (blood sodium concentration) will be made by 5 measurements carried out on the eve of the start and during the race, by microcapillary blood sample using the i-STAT technology and CHEM8+ cartridges.
Hydration saliva measurement | during 3 days of the race
  Hydration will be measured 5 times carried out on the eve of the start and during the race using saliva sample to measure the salivary osmolarity with the MX3 testing device.
Hydration by weight measurement | during 3 days of the race
  Weight in kg will be measured 5 times carried out on the eve of the start and during the race

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bouscaren, MD, Principal Investigator — Centre Hospitalier Universitaire de La REUNION
Locations (1):
- CHU Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouscaren N, Berly L, Descombes G, Tounkara B, Lacroix E, Lemarchand B, Racinais S, Millet GY. Thermoregulation and Hydration Dynamics in a 160-km Ultra-Endurance Race in a Tropical Environment: A Field Study on 80 Runners. Sports Med. 2025 Dec 4. doi: 10.1007/s40279-025-02356-6. Online ahead of print. PMID 41343039